CLINICAL TRIAL: NCT00002424
Title: A Multicenter, Double-Blind, Randomized Pilot Study to Compare the Safety and Activity of L-756423/Indinavir, 1600/800 Mg Qd or 800/400 Mg Bid Versus Indinavir, 800 Mg q8h, All in Combination With Stavudine and Lamivudine
Brief Title: A Study to Compare the Safety and Effectiveness of Indinavir Combined With Stavudine and Lamivudine
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 300B; 009-01; 009-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Drug Administration Schedule; Stavudine; HIV Protease Inhibitors; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — L 756423; Indinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: L-756423
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
This study will see how safe and effective against HIV the drugs L-756423 plus indinavir (IDV) are compared to just IDV when taken with stavudine (d4T) and lamivudine (3TC). The study will also see whether taking 1 large dose of L-756423/IDV once a day is as safe and effective as taking 2 smaller doses twice a day.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 4 treatment arms. In Group 1, patients receive a dose of L-756423/IDV once daily plus IDV placebo. In Group 3, patients receive a lower dose of L-756423/IDV twice daily (with the daily dosage equaling that of Group 1) plus IDV placebo. In Groups 2 and 4, patients receive equal dosages of IDV plus L-756423/IDV placebo. In all 4 groups L-756423 and IDV are blinded to the investigator and patient. All groups receive open-label d4T and 3TC. Patients routinely undergo a physical exam and have blood and urine tests to ensure the drugs' safety and tolerability, which will be evaluated by tabulation of adverse events and clinical assessment of laboratory data. In addition, CD4+ T cell and plasma viral RNA levels are measured to quantify the drugs' antiretroviral activity.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this trial if you:

* Have HIV infection.
* Have levels of CD4 cells of 100 cells/mm3 or greater.
* Have a viral load of 10,000 copies/ml or greater.
* Are 18 years of age or older.

Exclusion Criteria

You may not be eligible for this trial if you:

* Have ever taken anti-HIV drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - UCLA School of Medicine / Ctr for Research and Education, Los Angeles, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - ViRx / Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Associates in Research, Fort Myers, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Grady Mem Hosp, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Univ of Kentucky, Lexington, Kentucky
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Henry Ford Hosp, Detroit, Michigan
  - NYU Med Ctr / C & D Building, New York, New York
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York
  - SUNY at Stony Brook / Div of Infectious Disease, Stony Brook, New York
  - The Miriam Hosp, Providence, Rhode Island